CLINICAL TRIAL: NCT05576883
Title: Optimizing a Mobile Transdiagnostic Emotion Regulation Intervention for University Students: A Micro Randomized Trial
Brief Title: Optimization of a Mobile Transdiagnostic Emotion Regulation Intervention for University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus University Rotterdam (Other)
Responsible Party: Principal Investigator, Marilisa Boffo, Assistant Professor in Clinical Psychology and eHealth,, Erasmus University Rotterdam
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ETH2122-0677
Record Dates: First submitted 2022-10-06; First posted 2022-10-13 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Emotion Regulation; Stress; Depressive Symptoms; Anxiety
Keywords: Transdiagnostic intervention; Micro Randomized Trials; User research; Mental health; University Students
MeSH Terms: conditions — Emotional Regulation; Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study utilizes a Micro Randomized Trial [MRT] method to evaluate the effects of the intervention. Compared to a multi-arm trial, in which participants are randomized to an intervention or control group, in an MRT individuals are randomized repeatedly to different interventions during the trial which allows for a large number of observations of the targeted proximal outcome(s) per participant (in this case, emotional states). This design also allows us to investigate contextual moderators of proximal effects such as time of intervention delivery and emotional state.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emotion Regulation Intervention and Control Intervention (Other): Participants will be asked in the morning and in the evening at their self-selected time to evaluate their emotional state through ecological momentary assessment (EMA) and will be prompted to engage in an ER intervention (60% likelihood) or to read health information (40% likelihood). Upon completion they will evaluate the likability and helpfulness of the exercise or the article and re-evaluate their emotional state (post-EMA).
  The intervention consists of 20 ER exercises and 20 health facts. The ER intervention is based on different therapeutic approaches targeting various underlying transdiagnostic factors such as rumination, self-referential thoughts etc. The 20 health facts will act as a placebo intervention with no effect on emotion regulation and keep participants engaged in the post-EMA evaluation when they are not randomized to an exercise.
  The interventions and the control intervention materials were developed by the research team for the purposes of this study.
  Interventions: Behavioral: Transdiagnostic emotion regulation intervention

INTERVENTIONS:
Behavioral: Transdiagnostic emotion regulation intervention — The intervention under study includes 5 therapeutic approaches, namely: Positive psychology [PP], Mindfulness, Acceptance and Commitment Therapy [ACT], Breathing and relaxation, and Self-compassion [SC].
  The intervention consists of 4 core features:
  (i) monitoring through filling in EMAs assessing participants emotional states
  (ii) feedback through visualization of participant emotional states upon every completion of the EMAs
  (iii) exercises targeting different emotion regulation skills [i.e., upregulation of positive affect, mindfulness, cognitive defusion, breathing and relaxation, self-compassion) and health facts (i.e., control intervention) describing health information including nutrition, exercise, sleeping habits.
  (iv) psychoeducative articles describing the 5 therapeutic approaches (PP, ACT, Mindfulness, Breathing and Relaxation, SC)

SUMMARY:
This study will explore the functioning of a mobile transdiagnostic emotion regulation intervention designed for university students to optimize the uptake and the effectiveness of the intervention.

DETAILED DESCRIPTION:
It is estimated that globally between 12 and 50% of all university students are affected by mental health problems, the most common ones being anxiety, depression, and substance abuse. Over the past years online-based interventions have been spotlighted by researchers and clinicians as an avenue for a better outreach and provision of low threshold interventions aimed at primary and secondary prevention of mental health problems among the university students population.

As part of a student wellbeing program at the Erasmus University Rotterdam (EUR), a transdiagnostic mobile intervention consisting of a suite of preventative self-guided tools is being developed. Its' goal is to help students better manage their mental health by teaching them adaptive emotional regulation strategies.

The intervention includes exercises from different therapeutic approaches, and targets transdiagnostic factors such as negative self-referential thoughts, rumination, experiences of prolonged negative emotional states, and mental health literacy. The intervention is delivered via a smartphone and consists of 20 therapeutic exercises teaching students strategies like upregulation of positive affect, staying present in the moment, cognitive defusion, relaxation and breathing techniques, and self compassion skills.

The main goals of the study are to evaluate whether the intervention and its components have the intended effects on student's emotional states as well as get insight into students' engagement patterns and experience with the intervention. This will be done by utilizing an explanatory sequential mixed methods approach combining novel methods of online-intervention assessment, specifically Micro Randomized Trials (MRT) with semi-structured interviews, which will provide information on the lived experiences of the participants with the intervention and provide explanation of the quantitative results. The results of this trial will support the optimization and further development of the mobile application that will later be evaluated for its full-scale effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent
* Currently enrolled as a student at the Erasmus University Rotterdam
* Own a smartphone with an active phone number
* Feel comfortable speaking and writing in the English language
* Having a score between 5 (mild) and 19 (moderately severe) on the PHQ-9

Exclusion Criteria:

Participants are not eligible for this study if they:

* Experience significant suicidal thoughts over the past month
* Have a medical diagnosis of psychosis or bipolar disorder, severe clinical depression or anxiety disorder
* Are undergoing psychopharmacological treatment or treatment with experimental drugs

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Changes in a momentary emotional state | Day 2 - day 22
  Participants will be asked to evaluate seven emotional states before and after engaging in the ER intervention or control intervention by answering the question: "How [affect (e.g., happy)] do you feel at the moment?" Each of 7 emotional states is evaluated on a scale from 1 [Not at all] to 5 [Extremely]. The emotional states are combined into 2 categories of affect: negative (stressed, frustrated, sad, fatigued) and positive (happy, energetic, relaxed).
  Changes in the momentary emotional states (i.e., positive and negative affect) will be evaluated by looking at the responses on the pre and post EMA in the relation to whether a participant received an ER intervention or health information.
Changes in thought believability and discomfort after engaging in CD exercise | Day 2 - day 22
  When randomized to CD exercise, participants will be asked to evaluate their self-selected unhelpful thought answering the following questions on a scale from 1 (not at all uncomfortable/believable) to 100 (extremely uncomfortable / believable) before and after the exercise:
  "How uncomfortable is the thought?" "How believable (true) is the thought?"
  The effects of CD exercises will be assessed by comparing the pre and post scores on the two thought parameters.
Objective engagement patterns: Engagement metrics | Day 2 - day 22
  Objective engagement patterns with the intervention will be assessed using descriptive statistics of engagement metrics (i.e., exercise completion rates, average time spent, and times of the day where participants completed the exercises) per exercise and exercise category. In addition, a correlational analysis will be used to evaluate whether there is a relationship between time of the day and exercise completion rates.
Objective engagement patterns: Relationship between time of the day and exercise completion | Day 2 - day 22
  A correlational analysis will be used to evaluate whether there is a relationship between the time of the day participants engaged in an exercise and exercise completion rates.
Subjective engagement patterns: Exercise likeability and helpfulness | Day 2 - day 22
  Subjective engagement patterns will be evaluated by combining exercise likeability and helpfulness ratings with information from the semi-structured interviews.
  Exercise likeability and helpfulness are assessed with items rated on a scale from 1 (not at all) to 5 (very much):
  "How much did you like the exercise?" "How helpful did you find the exercise?"
Subjective engagement patterns: User experience | Up to 3 weeks upon completion of the Micro Randomized Trial
  Semi-structured interviews will be conducted with a subsample of participants (n=21) within three weeks upon completion of the MRT. University students will be asked to report on their general experience with intervention as well as intervention categories and separate exercises. Example questions are: "What do you think about the intervention?", "What kind of difficulties did you experience while using it?",

SECONDARY OUTCOMES:
Changes in ER skills | At the baseline and day 23
  ER skills will be measured with the Emotion Regulation Skills Questionnaire [ERSQ] that evaluates seven types of ER skills: awareness, sensation, clarity, understanding, acceptance, tolerance, compassionate self-support, readiness to confront distressing situations, and modification of negative emotions. The 27 items are rated on a scale from 0 [ not at all ] to 4 [ almost always ]. Higher scores on the ERSQ subscales and the overall ERSQ score indicate higher ER skills.
Changes in Anxiety symptoms | At the baseline and day 23
  Symptoms of anxiety will be measured with the Generalized Anxiety Disorder questionnaire [GAD-7] Participants will indicate how often they have been bothered by different symptoms over the last two weeks on a scale from 0 (not at all) to 3 (nearly every day). The summed scores for GAD-7 range between 0-21, with higher scores indicating higher levels of depression and anxiety symptoms
Changes in Depressive symptoms | At the baseline and day 23
  Symptoms of depression will be measured with the Patient Health Questionnaire [PHQ-9]. Participants will indicate how often they have been bothered by different symptoms over the last two weeks on a scale from 0 (not at all) to 3 (nearly every day). The summed scores for PHQ range from 0-27, with higher scores indicating higher levels of depression and anxiety symptoms
Changes in stress levels | At the baseline and day 23
  Perceived Stress Scale [PSS-10] will be used to assess stress levels. Participants will be asked to indicate how often they felt or thought a certain way over the last month on a scale from 0 [never] to 5 [very often]. The summed score ranges from 0 - 40, with higher scores indicating higher levels of perceived stress symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus University Rotterdam, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data [and code] produced in the project will be shared in a research data repository [EUR Data Repository (EDR) and Open Science Framework (OSF)]. A DCMI [Dublin Core Metadata Initiative] standard will be used to document this research. There will be a temporary restriction on re-using of the data (Embargo period of 6 months).
  Data [and code] that will be shared in a research data repository are: Anonymized survey data, Codebook and Blank Questionnaires, Readme text file (general description of the data, including date of collection, selection procedure of participants, tools used to collect the data etc.), and scripts of data analysis.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The data will come available after the embargo period of 6 months.

REFERENCES:
- [Background] Laure T, Engels RCME, Remmerswaal D, Spruijt-Metz D, Konigorski S, Boffo M. Optimization of a Transdiagnostic Mobile Emotion Regulation Intervention for University Students: Protocol for a Microrandomized Trial. JMIR Res Protoc. 2023 Oct 27;12:e46603. doi: 10.2196/46603. PMID 37889525
- See also: Study Pre-print — http://psyarxiv.com/xgq2r/